CLINICAL TRIAL: NCT02778906
Title: Abatacept Reversing Subclinical Inflammation as Measured by MRI in ACPA Positive Arthralgia (ARIAA)
Brief Title: Abatacept Reversing Subclinical Inflammation as Measured by MRI in ACPA Positive Arthralgia
Acronym: ARIAA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-477
Record Dates: First submitted 2015-02-02; First posted 2016-05-20 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Arthralgia; Arthritis
Keywords: Abatacept
MeSH Terms: conditions — Arthralgia; Arthritis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abatacept (Active Comparator): Abatacept 125 mg s.c. weekly
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): Placebo (NaCl 0,9%) s.c. weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept — Administration of Abatacept s.c. 125mg/weekly according to the Label for Rheumatoid arthritis
  Other Names: Orencia
  Arms: Abatacept
Drug: Placebo — Administration of the comparator s.c. weekly in comparable to verum
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
This is a randomised double-blinded placebo-controlled multi centre study in 98 patients with ACPA positive arthralgia. The study is composed of 2 arms with a 1:1 randomisation at baseline: Treatment phase will be 6 months. Group 1: Abatacept s.c. 125 mg weekly for 6 months vs. Group 2: Placebo s.c. for 6 months. After 6 months both groups will run into the follow up period for another 12 months up to month 18. Patients developing arthritis will be treated according to local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Females and males aged ≥ 18 years at time of consent
* ACPA (with or without RF)
* Joint pain (hand, feet, knee, shoulder or elbow) present for at least 6 weeks prior to inclusion or in past history
* Presence of synovitis (synovialitis or tenosynovitis) or osteitis in MRI of the dominant hand at baseline
* Women of childbearing potential or men capable of fathering children must be using effective contraception during treatment with abatacept and up to 14 weeks after the last dose of abatacept treatment.
* Must understand and voluntarily sign an informed consent form including written consent for data protection
* Must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Presence of arthritis in hand, feet, knee, shoulder or elbow joints defined as swelling
* Current treatment with glucocorticoids conventional or biologic DMARDs
* Previous treatment with abatacept
* Investigational study drug within 4 weeks (or 5 half lives, whichever is longer) prior to randomization
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Any other autoimmune or inflammatory disease such as SLE, PSS, MCTD, SpA, Behcet disease, vasculitis or autoimmune hepatitis.
* Any malignancy in the last 5 years
* Chronic infection such as latent TB (TB not adequately treated according to guidelines) or hepatitis B or C infection
* Immunocompromised or HIV-positive patients
* Uncontrolled severe concomitant disease
* Patients who are younger than 18 years or are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (according to § 40 Abs. 4 and § 41 Abs. 2 and Abs. 3 AMG).
* Pregnant or lactating females
* Patients who possibly are dependent on the Principal Investigator or Investigator (e.g. family members).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an improvement of acute inflammation characterised as improvement of synovitis (synovialitis or tenosynovitis) or osteitis in the MRI of the dominant hand after 6 months of treatment with abatacept or placebo | 6 months

SECONDARY OUTCOMES:
RAMRIS synovitis score in the dominant hand 12 and 18 months. | 6,12,18 months
Tenosynovitis score in the dominant hand. | 6,12,18 months
Proportion of patients with new or persistent arthralgia. | 6,12,18 months
Time to disappearance of arthralgia. | 6 months
Proportion of patients with clinical arthritis defined by joint swelling | 6,12,18 months
Proportion of patients with RA (ACR/EULAR 2010 criteria) | 6,12,18 months
Proportion of patients with radiological progress in HR-pQCT analysis comparing baseline image with end of study image. | 18 months
Tender Joint Count 68 | 3,6,9,12,15 and 18 months
Disease activity score (DAS) 28 | 3,6,9,12,15 and 18 months
Visual analogue scale (VAS) pain | 3,6,9,12,15 and 18 months
Duration of joint stiffness | 3,6,9,12,15 and 18 months
Health assessment Questionnaire (HAQ-DI) | 6,12 and 18 months
Rheumatoid Arthritis Impact of Disease (RAID) | 6,12 and 18 months
Short Form 36 (SF-36) | 6,12 and 18 months
Bone mineral density (BMD) | 18 months
Bone volume per tissue volume (BV/TV) | 18 months
Cortical width in the micro-CT of the distal radius | 18 months
Cortical porosity in the micro-CT of the distal radius | 18 months
RAMRIS erosion score in the dominant hand 12 and 18 months. | 6. 12. 18 months
RAMRIS osteitis score in the dominant hand 12 and 18 months. | 6,12,18 months
Swollen Joint Count 68 | 3,6,9,12,15 and 18 months
Visual analogue scale (VAS) patient global | 3,6,9,12,15 and 18 months
Visual analogue scale (VAS) physician global | 3,6,9,12,15 and 18 months
Cortical width in the micro-CT of the metacarpal heads | 18 months
Cortical porosity in the micro-CT of the metacarpal heads | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schett, Prof. Dr. univ., Principal Investigator — University Clinic Erlangen, Department of Internal Medicine 3, Rheumatology & Immunology
Locations (9):
- Germany (9):
  - Klinikum Bad Abbach, Bad Abbach
  - Charite Berlin, Berlin
  - Praxis für Rheumatologie und Innere Medizin, Berlin
  - Clinic Burghausen, Burghausen
  - Krankenhaus Porz Am Rhein, Cologne
  - University Clinic Erlangen, Erlangen
  - Centrum für innovative Diagnostik und Therapie (Ciri) Rheumatologie/Immunologie, Frankfurt
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Rheumazentrum Ruhrgebiet, Herne

IPD SHARING:
Plan to Share IPD: No